CLINICAL TRIAL: NCT05802160
Title: A Good Start Matters for Parents and Children: an MHealth Parenting Intervention to Promote a Healthy Child Development
Brief Title: The Good Start Matters - Parenting Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Louise Masse, Professor, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H18-01434(2)
Record Dates: First submitted 2023-03-15; First posted 2023-04-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-05

CONDITIONS: Parenting Practices; Co-parenting Practices; Child Eating and Dietary Behaviors; Child Physical Activity/active Play/outdoor Play; Child Screen Time
Keywords: Parenting intervention; mHealth; parenting practices; co-parenting; eating behavior; physical activity; active play; screen time
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Good Start Matters Parenting intervention (Experimental): The intervention group will receive immediate access to the app where the Good Start Matters - Parenting intervention will be delivered over a 2-months period.
  Interventions: Behavioral: Good Start Matters - Parenting intervention
- Control (No Intervention): The control group will not receive access to the intervention until they complete the follow-up measures (after 10 weeks).

INTERVENTIONS:
Behavioral: Good Start Matters - Parenting intervention — The Good Start Matters - Parenting intervention is a 2-month mobile-Health (mHealth) parenting program that aims to improve parenting practices and child health behaviors among British Columbian families of preschoolers. This intervention uses a familial approach and blends the best practices and evidence to promote positive parenting regarding 3 main areas: nutrition, physical activity, and screen-time; which altogether aim to support the development of healthy habits among young children. The mHealth app releases new material on a weekly basis and participants' engagement with the app takes about 30 minutes per week.
  Arms: Good Start Matters Parenting intervention

SUMMARY:
Early childhood is an important period where the family can support the development and maintenance of healthy eating and active behaviors to prevent or reduce childhood obesity. With this ultimate goal, we designed the Good Start Matters - Parenting program, which aims to engage families in positive parenting practices that support healthy child behaviors, and aim to evaluate the efficacy of this intervention with a Randomized Controlled Trial (RCT). The Good Start Matters - Parenting program is a 2-month mobile-Health (mHealth) parenting intervention which promote positive parenting (primary outcome) and support children's healthy nutrition, physical activity, and decrease screen-time (secondary outcomes).

DETAILED DESCRIPTION:
Early childhood is an important learning period where dietary, physical activity and sedentary habits are forming, and developing unhealthy habits will set children up for obesity and other health risks later in life. Moreover, during early childhood the familial environment plays a key role in shaping children's behaviors through their parenting practices, which altogether illustrate the potential of the early years as a developmental period with opportunities for obesity prevention. This Randomized Controlled Trial (RCT) evaluates the efficacy of the Good Start Matters - Parenting intervention, a mobile-Health (mHealth) aimed at improving parenting and co-parenting practices and child health behaviors among British Columbian families of preschoolers. Participating families complete measurement tools at baseline and after 10 weeks. Families randomized into the intervention condition receive immediate access to the app, and control families receive access to the app after the completion of the second assessment. We expect that compared to control group families, intervention group families significantly improve their parenting and co-parenting practices and improve child health behaviors after 2 months of app use.

ELIGIBILITY:
Inclusion Criteria:

Children must be:

* Attending a childcare center invited to participate in the Good Start Matters study.
* Older than 2.5 and younger than 6 years

Parents must:

* Be the primary caregiver/legal guardian of an eligible child OR share childrearing responsibilities with an already enrolled primary caregiver/legal guardian of an eligible child
* Be fluent in English
* Have a cellphone number and smartphone device where they can receive text messages and download and access the app

Exclusion Criteria:

Parents and children:

- Currently participating in a pediatric weight management program or in a nutritional program are not eligible.

Children:

* With severe dietary restrictions that limit their ability to follow general nutritional guidelines for toddlers and preschoolers are not eligible.
* With severe physical limitations that limit their ability to follow general movement behavior guidelines for toddlers and preschoolers are not eligible.

Ages: 30 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Change in Parenting practices (parent outcome) | Two time points (baseline and 10 weeks post intervention)
  Questions adapted from the "Food and Physical Activity Item Banks" (Masse et al 2020) to specifically assess parenting practices related to food, physical activity and screen time. The scale ranges from 1-5 in most items, and higher scores indicate greater endorsement of each parenting practice.

SECONDARY OUTCOMES:
Change in Co-Parenting practices (parent outcome) | Two time points (baseline and 10 weeks post intervention)
  Questions adapted from the "Coparenting Relationship Scale" from Feinberg et al (2012) to measure co-parenting agreement specifically regarding the child eating and movement behaviors. The scale ranges from 1-4 and all items will be coded in the same direction to have greater scores representing greater coparenting agreement.
Change in Eating and dietary behaviors (child outcome) | Two time points (baseline and 10 weeks post intervention)
  Questions from the "Children´s Eating Behaviors Questionnaire" (CEBQ) (Wardle et al, 2001), questions based on "Canada´s Food Guide" recommendations, and questions created for the current study to assess a variety of children´s eating behaviors around food (e.g., fussiness, emotional overeating) and intake of key food markers (e.g., vegetables, fruits, sugary drinks). Specifically for the CEBQ scale, response options range from 1-5, and all items will be recoded in the same direction to have greater scores representing greater frequency of each child behavior.
Change in Physical activity (child outcome) | Two time points (baseline and 10 weeks post intervention)
  Questions adapted from Burdette et al. (2004) to examine child physical activity through active play and outdoor play. Greater scores indicate greater active play and outdoor play time.
Change in Screen time (child outcome) | Two time points (baseline and 10 weeks post intervention)
  Questions created for this study to examine children's time in front of screens. Greater scores indicate greater screen time.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Masse, PhD, Principal Investigator — University Of British Columbia & BC Children's Hospital Research Institute
Locations (1):
- University of British Columbia / BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De-Jongh Gonzalez O, Tugault-Lafleur CN, Mah JWT, Masse LC. The Good Start Matters mHealth Parenting Program: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 23;14:e72642. doi: 10.2196/72642. PMID 41129815